CLINICAL TRIAL: NCT05063409
Title: A Randomized Prospective Trial of Fresh Frozen Plasma (FFP) to Packed Red Blood Cell (PRBC) Ratio: Comparison of a Traditional (1:4) to Liberal (1:1)FFP Transfusion Policy During Burn Excision and Grafting
Brief Title: Transfusion Ratio of Fresh Frozen Plasma (FFP) to Packed Red Blood Cell (PRBC) During Burn Excision and Grafting
Acronym: FFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Tina L Palmieri, Assistant Chief of Burns, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHC 70014; 216586 (Other: UC Davis IRB)
Record Dates: First submitted 2012-08-31; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Burn Injury
Keywords: FFP; PRBC; Burn
MeSH Terms: conditions — Burns | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:1 Ratio of FFP to PRBC (Active Comparator): Randomized treatment to receive blood products at a ratio of 1:1 FFP to PRBC during the operative period (start of surgery to 12 hours post operatively)
  Interventions: Other: Treatment
- 1:4 Ratio FFP to PRBC (Active Comparator): Randomized treatment to receive blood products at a ratio of 1:4 FFP to PRBC during the operative period (start of surgery to 12 hours post operatively)
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Blood product transfusion at a ratio of 1:1 FFP to PRBC or 1:4 FFP to PRBC during the operative period (start of surgery to 12 hours post operatively)

SUMMARY:
The purpose of this study is to determine if burn injured patients who receive blood transfusions in the operating room have better outcomes when given transfusions at a set ratio (1:1)of PRBC to FFP.

Traditionally, patients that need blood transfusions during surgery are given mostly packed red blood cells (PRBC) and some fresh frozen plasma (FFP). This is usually about 1:4 ratio of FFP to PRBC.

In this study, we will compare this traditional approach (1:4) to a 1:1 ratio of FFP to PRBC during the operative period.

The hypothesis of the study is that the use of FFP/PRBC ratio of 1:1, compared to a ratio of 1:4 will result in a(n)

1. decrease in the amount of blood transfused in the operating room
2. decrease in the amount of blood transfused during hospitalization
3. improvement in coagulation parameters (PT/PTT, INR, antithrombin III, Protein C and Fibrinogen in the operative period (from operation start to 12 hours post operatively) and at 24 hours postoperatively
4. decrease the hospital length of stay, lung dysfunction, infections, and mortality

DETAILED DESCRIPTION:
The hypothesis of the study is that the use of a fresh frozen plasma/packed red blood cells (FFP/PRBC) ratio of 1:1, compared to a ratio of 1:4 during operative excision of >20% TBSA will: result in a decrease in the amount of blood transfused in the operating room, a decrease in the amount of blood transfused during hospitalization, an improvement in coagulation parameters (PT/PTT, INR) in the operative period (from operation start to 12 hours postoperatively) and at 24 hours postoperatively, and a decrease in hospital length of stay, lung dysfunction, number of infections, and mortality.

The primary objective of the study is to determine if aggressive correction of intraoperative coagulopathy during burn excision and grafting results in improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 1 month to </= 18 yrs of age
* Admitted to Shriners Hospitals for Children Northern California
* Patient has a third degree burn >/= 20 % total body surface area (TBSA)

Exclusion Criteria:

* Infants < 5 kg
* Pregnancy

  * 18 years of age
* Inability or unwillingness to receive blood products
* Pre-existing need for hemodialysis
* Brain death or imminent brain death
* Non-survivable burn as determined by the attending burn surgeon
* Pre-existing hematologic disease
* Closed head injury with Glasgow Coma Score <9

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
change in the amount of blood transfused in the operating room and during hospitalization | Baseline to 12 months- From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  All transfusions during the operative period and entire hospitalization will be documented

SECONDARY OUTCOMES:
change in rate of survival | From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  survival outcome as captured at discharge
change in coagulopathy in the operative period as defined by change in PT/PTT measurement | from operation start to 12 hours post operatively
  PT/PTT obtained pre and post operatively per protocol
change in hospital length of stay | From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  Number of days in hospital from admit to discharge
change in number of infectious episodes | From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  number of new onset infections captured as defined by the Burn Sepsis Consensus Conference
change in organ dysfunction | From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  Change in organ dysfunction as evidenced by change in MODS
change in pulmonary dysfunction | From date of hospital admit to date of hospital discharge, assessed over duration of hospitalization up to 12 months
  pulmonary dysfunction measured by P:F ratio and number of days on mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Tina Palmieri, MD, Principal Investigator — SHCNC and UC Davis
Locations (1):
- Shriners Hospital for Children Northern California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmieri TL, Sen S, Falwell K, Greenhalgh DG. Blood product transfusion: does location make a difference? J Burn Care Res. 2011 Jan-Feb;32(1):61-5. doi: 10.1097/BCR.0b013e318204b3ea. PMID 21107270